CLINICAL TRIAL: NCT06135961
Title: Implementation of Intrapartum Non-invasive Electrophysiological Monitoring
Brief Title: Intrapartum Non-invasive Electrophysiological Monitoring
Acronym: NIEM-II
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maxima Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, Phebe Berben, Medical doctor, PhD Candidate, Coordinating Investigator NIEM-II study, Maxima Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: NL82822.015.22
Record Dates: First submitted 2023-11-02; First posted 2023-11-18 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Fetal Monitoring; Non-invasive; Cardiotocography; Electrocardiography; Caesarean Section

STUDY DESIGN:
Intervention Model Description: Eligible women will be prospectively included in the cohort receiving conventional CTG monitoring. From the eligible women in the prospective cohort a random sample (90.9%) will be offered eCTG monitoring via a computer generated random collection. Participants will receive eCTG monitoring from the start of fetal monitoring during labour until 1.5 hour after delivery. A retrospective cohort of 2100 women who received conventional CTG monitoring between April 2019 and February 2023 will be added to the prospective cohort for statistical analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- eCTG monitoring (Active Comparator): eCTG monitoring with the Nemo Fetal Monitoring System (Nemo Healthcare B.V., Veldhoven, the Netherlands).
  The NFMS consists of a wireless and beltless electrode patch on the maternal abdomen. It monitors fetal heart rate by fetal electrocardiography, maternal heart rate by maternal electrocardiography and the electrical activity of the uterine muscle by electrohysterography.
  The advantage of the NFMS is that it is a safe method that can be used in all situations that are contraindicated for invasive monitoring. Furthermore, it can be used when the membranes are not ruptured and the patch does not have to be repetitively repositioned during labor. Because the NFMS is wireless, it gives women more freedom of movement during labor.
  Interventions: Device: eCTG monitoring with the NFMS
- Conventional CTG monitoring (No Intervention): Philips Avalon FM 30 (Philips Healthcare, Eindhoven, the Netherlands).
  The fetal heart rate is measured non-invasively by doppler ultrasound or invasively by fetal scalp electrode. The uterine activity and maternal heart rate is measured by tocodynamometry.

INTERVENTIONS:
Device: eCTG monitoring with the NFMS — Device: Nemo Fetal Monitoring System (Nemo Healthcare B.V., Veldhoven, the Netherlands)
  Arms: eCTG monitoring

SUMMARY:
Conventional cardiotocography (CTG) has been used extensively for more than 50 years to monitor the fetal condition during labour, but since the rate of operative deliveries keeps rising, its ability to improve neonatal outcomes is unsatisfactory. A transabdominal non-invasive and wireless alternative which overcomes the shortcomings of conventional methods is electrophysiological CTG (eCTG) monitoring. In eCTG the fetal heart rate (FHR) is measured by fetal electrocardiography (NI-fECG) and uterine activity (UA) by electrohysterography (EHG). Both NI-fECG and EHG have been proven more accurate and reliable than conventional non-invasive methods and are less affected by maternal body mass index (BMI).

This study aims to evaluate the mode of delivery, maternal and perinatal outcomes, costs and patient and healthcare professionals perspectives on eCTG monitoring versus the conventional CTG during labour at term with a singleton fetus in cephalic position.

The eCTG provides a more accurate assessment of the fetus and the UA, compared to the conventional CTG. This allows for optimization of the contraction pattern during high-risk deliveries. We hypothesize that this will reduce the number of operative interventions and improves perinatal outcome. There are three reasons why an improvement in the contraction pattern by the eCTG can influence our outcomes:

1. EHG can detect excessive UA more accurately. Increased UA is a major risk for fetal distress. In this case, stimulation with oxytocin should be reduced or stopped. More adequate interpretation of FHR, reduced tachysystole and reduced hypertonia is expected to result in fewer instrumented vaginal deliveries and a reduction of caesarean sections due to fetal distress.
2. EHG can demonstrate unorganized UA that needs to be corrected with a higher dose of oxytocin to enhance contraction frequency and efficiency. This can result in a less exhausted uterine muscle, shorter time to delivery, less vacuum deliveries and caesarean sections due to failure of progress. A shorter time to delivery will also result in a reduction of infections and blood loss.
3. Accurate registration of the relation between the contraction and decelerations of FHR, is expected to result in more reliable assessment of the fetal condition. This can result in fewer unnecessary operative deliveries and less unpredictable poor perinatal outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Minimal age of 18 years old
* Pregnant women with a gestational age between 37+0 and 42+0 weeks and days
* Indication for fetal monitoring during labour
* Singleton fetus in cephalic position
* Oral and written informed consent is obtained

Exclusion Criteria:

* Insufficient knowledge of Dutch or English language
* Women with a multiple pregnancy
* Fetal and/or maternal cardiac arrhythmias
* Contraindications to abdominal patch placement (dermatologic diseases of the abdomen precluding preparation of the abdomen with abrasive paper)
* Women connected to an external or implanted electrical stimulator, such as Transcutaneous Electro Neuro Stimulation (TENS) and pacemaker (because of disturbance of the electrophysiological signal)
* Women who take a bath for multiple times during delivery and/or who take a bath for > 1 hour during the first stage of labour and/or who take a bath in the second stage of labour. eCTG monitoring is impossible in bath because the Bluetooth signal is disturbed. In bath, monitoring will be performed by conventional CTG monitoring. However, it is possible to take a shower with eCTG monitoring
* Treatment plan (with intervention plan) already made before inclusion is completed.
* Women who were included in the study, but when circumstances before labour call for delivery of the baby by unplanned caesarean section.
* There is insufficient time for proper counselling
* Women admitted with a clinical diagnosis of sepsis with hypotension (i.e. septic shock).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3471 (Estimated)
Dates: Start 2023-11-20 (Actual); Primary Completion 2025-11-20 (Estimated); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
The number of operative interventions during labor | During delivery
  cesarean section or instrumental vaginal delivery

SECONDARY OUTCOMES:
Duration of the first stage of labor in minutes | 0-10 cm dilation during labor
Duration of the second stage of labor in minutes | Start pushing until childbirth
The timing and reason of operative interventions during labor | During delivery
  Timing is defined as:
  * The decision delivery interval for the intervention: emergency ('code red' or within <30 minutes of the decision) or ≥ 1 hour
  * As the phase of delivery: first stage or second stage of labor
The number of participants with analgesia for pain reduction: epidural or/and remifentanil | During delivery
Perineal laceration (grade 1, 2, 3a, 3b, 3c, 4) | Directly after childbirth
The number of participants with a mediolateral episiotomy and reason for the episiotomy | Directly after childbirth
Number (percentage) and result of fetal blood sampling during the primary and secondary stages of labour | During delivery
Perinatal mortality | During pregnancy up to seven completed days of life
  Perinatal mortality is defined as the number of fetal deaths past 22 completed weeks (154 days) of gestation plus the number of deaths among live-born children up to seven completed days of life
Neonatal mortality | After the seventh day but before the 28th day of life
  Neonatal mortality is defined as the number of neonatal deaths after the seventh day but before the 28th day of life
The number of neonates with hypoxic ischemic encephalopathy | childbirth - 28th day postpartum
The number of neonates with Neonatal Respiratory Distress Syndrome (RDS) | childbirth - 28th day postpartum
The number of neonates with Meconium Aspiration Syndrome (MAS) | childbirth - 28th day postpartum
The number of neonates with convulsions | childbirth - 28th day postpartum
The number of neonates with Clinical early onset sepsis | childbirth - 28th day postpartum
  Clinical early onset is defined as clinical sepsis within the first 72 hours after birth with > 3 days of antibiotics
The number of neonates with Confirmed early onset sepsis | childbirth - 72 hours after childbirth
  Confirmed early onset sepsis is defined as positive cultures of blood, cerebrospinal fluid, or urine from the first 72 hours after birth
The number of neonates with admission to Neonatal Intensive Care Unit | childbirth - 28th day postpartum
Length of Admission to Neonatal Intensive Care Unit | childbirth - 28th day postpartum
  In days
Reason for the admission to Neonatal Intensive Care Unit | childbirth - 28th day postpartum
The number of neonates with the need for mechanical ventilation | childbirth - 72 hours after childbirth
  The number of neonates with the need for mechanical ventilation within the first 72 hours after birth
The number of neonates with a 5 minute Apgar score <7 | 5 minutes after childbirth
The number of neonates with a neonatal acidosis at birth | Directly after childbirth
  It is defined as cord artery pH < 7.05 and base deficit > 12 mmol/L directly after birth. The definition is set as pH < 7.10 and base deficit > 12 mmol/L in cases with only an umbilical vein sample (one available blood gas sample or the pH difference between two samples below 0.03)
Maternal mortality | During pregnancy and childbirth or within 42 days of termination of pregnancy
  Maternal mortality or 'pregnancy-related death' is defined as death from any cause related to or aggravated by the pregnancy or its management (excluding accidental or incidental causes) during pregnancy and childbirth or within 42 days of termination of pregnancy, irrespective of the duration and site of the pregnancy
The number of mothers admitted to the Intensive Care Unit | childbirth until six weeks postpartum
The number of mothers with a thromboembolic event | childbirth until six weeks postpartum
The number of mothers with an uterine rupture | childbirth until six weeks postpartum
The number of mothers with an obstetric haemorrhage | childbirth until 24 hours after childbirth
  Obstetric haemorrhage > 1000 millilitres within 24 hours after giving birth
The number of mothers with a postpartum anemia due to postpartum haemorrhage with requires red cell transfusion | childbirth until six weeks postpartum
The number of mothers with a suspected or confirmed postpartum infection requiring antibiotics | childbirth until six weeks postpartum
  i.e. chorioamnionitis, endometritis, wound infection and/or urinary tract infection.
Patient satisfaction by questionnaires | 2-6 hours after childbirth
  Validated Birth-Satisfaction-Scale-Revised questionnaire and a non-validated questionnaire.
Professional satisfaction by questionnaire | 1 year after the start of the study
  Non-validated questionnaire
Costs as a business case model until six weeks postpartum | Delivery until six weeks postpartum
For eCTG monitoring: amount of signal loss in percentage of total duration during labour | During delivery
  The amount of signal loss will be calculated based on the CTG. Signal loss is defined as minutes without registration of the fetal heart rate
For eCTG monitoring: frequency of switch from Nemo Fetal Monitoring System to conventional CTG + reason, timing and success percentage of the switch | During delivery
For eCTG monitoring: EHG pattern within the first 1.5 hours postpartum and the possible association with the amount of bloodloss, medication use and time to placental expulsion | First 1.5 hours postpartum
For eCTG monitoring: EHG pattern before and after labour analgesia and the possible association of EHG pattern with labour analgesia | During delivery

CONTACTS AND LOCATIONS:
Locations (1):
- Maxima MC, Veldhoven, North Brabant, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication

REFERENCES:
- [Derived] Berben PBQ, de Klerk ND, van der Ven M, Fransen AF, Niemarkt HJ, van den Heuvel ER, van der Hout-van der Jagt MB, Oei SG, van Laar JOEH. Non-invasive electrophysiological monitoring vs conventional monitoring during labour in a tertiary obstetric care centre in the Netherlands: study protocol of a cohort intervention random sampling study (NIEM-II study). BMJ Open. 2025 Jul 22;15(7):e102901. doi: 10.1136/bmjopen-2025-102901. PMID 40701589